CLINICAL TRIAL: NCT00355719
Title: Clinical Pilot Trial to Evaluate the Influence of Nevirapine in Exposure to Atazanavir in Steady State Equilibrium in HIV-infected Adult Patients.
Brief Title: Study to Evaluate the Influence of Nevirapine to Atazanavir in Steady State Equilibrium in HIV Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Germans Trias i Pujol Hospital (Other)
Collaborators: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other); Hospital San Jaime de Calella (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEVIATAZ; 2006-001140-31
Record Dates: First submitted 2006-07-24; First posted 2006-07-25 (Estimated); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: HIV Infections
Keywords: Nevirapine; Atazanavir; Pharmacokinetics; Interactions
MeSH Terms: conditions — HIV Infections | interventions — Atazanavir Sulfate; Ritonavir; Nevirapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nevirapine-atazanavir (Experimental): Atazanavir/ritonavir 300/100 mg once daily for ≥2 weeks. Nevirapine was added at a dose of 200 mg once daily from days 0 to 14, and 200 mg twice daily from days 14 to 28.
  Interventions: Drug: Atazanavir (Reyataz); Drug: Ritonavir (Norvir); Drug: Nevirapine (Viramune)

INTERVENTIONS:
Drug: Atazanavir (Reyataz) — Atazanavir (Reyataz): capsules 150 mg (2 capsules/24h)
Drug: Ritonavir (Norvir) — Ritonavir (Norvir): capsules 100 mg (1 capsule/24h)
Drug: Nevirapine (Viramune) — Nevirapine (Viramune): tablets 200 mg (1 tablet/12h*)

SUMMARY:
The purpose of this study is to evaluate the influence of nevirapine in exposure to atazanavir boosted with ritonavir, in steady state equilibrium, in HIV-infected adult patients.

DETAILED DESCRIPTION:
In recent years, new treatment strategies have appeared aimed at reducing the risk of treatment-derived toxicity without compromising efficacy.

Of the recent antiretroviral drugs, atazanavir is a protease inhibitor (PI) whose pharmacokinetic profile allows it to be given in a single daily take with a scant impact on lipid metabolism. This second characteristic makes atazanavir a good alternative for patients with a high vascular risk. However, one of its drawbacks is that it may present clinically relevant interactions with other drugs.

Another antiretroviral agent with a scant impact on lipid metabolism is nevirapine. Different studies have described an improvement in lipid profile, as well as a less atherogenic tendency in patients treated with nevirapine. Moreover, the combination of nevirapine with PI drugs in the context of nucleoside-sparing strategies may permit a suitable control of viral replication, and an improvement in the mitochondrial toxicity derived from treatment with NTRI, which may possibly result in a minor incidence or in a clinical improvement of lipodystrophy.

The combination of atazanavir with nevirapine may be of major interest in HIV-infected patients that have had a cardiovascular event (secondary prevention) or are at a high risk of having one (primary prevention). Similarly, this combination of drugs may be promising as a nucleoside-sparing strategy. However, according to preliminary data, the joint administration of nevirapine with atazanavir may lead to a reduction in the atazanavir plasma concentration. Thus, before evaluating the clinical utility of this combination of drugs, pharmacokinetic studies evaluating the existence of significant pharmacokinetic interactions between both are necessary

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years.
* Patients infected by HIV-1 (at least one documented positive Western-Blot).
* Stable antiretroviral treatment with atazanavir boosted with ritonavir (300/100 mg QD) for at least 14 days.
* Absence of acute infections and/or tumours in the three months prior to inclusion.
* Subject able to follow the treatment period.
* Transaminase values (AST/ALT) below 5 times the upper limit of the interval of normality.
* In women, negative pregnancy test or not of fertile age (defined as at least one year from menopause or undergoing any surgical sterilisation technique), or undertaking to use a barrier contraceptive method during the study.
* Signature of the informed consent.
* Undetectable viral load.

Exclusion Criteria:

* Failure to comply with any of the inclusion criteria.
* Record of allergic hypersensitivity or intolerance to the investigational medication.
* Any clinical or historic observation that might interfere in the pharmacokinetics of the medication, such as gastrointestinal diseases or surgery (except herniotomy or appendectomy), alterations in the composition of plasma proteins, any indication of hepatic or renal dysfunction.
* Patients that have been given tenofovir, omeprazole or other proton pump inhibitors or any other medication with relevant interactions with atazanavir within the two weeks prior to the screening visit.
* Active consumption of alcohol (> 50 g/day) or illegal drugs (except cannabis).
* Suspicion of unsuitable antiretroviral treatment compliance.
* Pregnancy or breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-01; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of the study will be the atazanavir plasma concentration | at baseline and week 4

SECONDARY OUTCOMES:
Proportion of patients with atazanavir plasma concentrations < 0.15 mg/L | at baseline and week 4
Proportion of patients with nevirapine plasma concentrations > 6.0 mg/L | at baseline and week 4
Incidence of adverse events and anomalies in the laboratory tests (haemogram, AST / ALT / FA / GGT, bilirubin, creatinine, urea). | during the 8 weeks of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Bonaventura Clotet, MD,PhD, Principal Investigator — LLuita contra la Sida Foundation-HIV Unit; Jose Molto, MD,PhD, Principal Investigator — LLuita contra la Sida Foundation-HIV Unitat; Josep Mª LLibre, MD,PhD, Principal Investigator — Lluita contra la Sida Foundation- HIV Unit; Sílvia Valero, Principal Investigator — Hospital Sant Jaume de Calella
Locations (2):
- Spain (2):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Sant Jaume de Calella, Calella, Barcelona